CLINICAL TRIAL: NCT06401577
Title: Diabetes RElated to Acute Pancreatitis and Its Mechanisms: Metabolic Outcomes Using Novel CGM Metrics (DREAM-ON) - An Observational Cohort Study From the Type 1 Diabetes in Acute Pancreatitis Consortium (T1DAPC)
Brief Title: Diabetes RElated to Acute Pancreatitis and Its Mechanisms: Metabolic Outcomes Using Novel CGM Metrics
Acronym: DREAM-ON
Status: Recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Benaroya Research Institute (Other); Cedars-Sinai Medical Center (Other); University of Southern California (Other); Indiana University (Other); Johns Hopkins University (Other); Ohio State University (Other); Stanford University (Other); University of Florida (Other); AdventHealth (Other); University of Illinois at Chicago (Other); Northwestern University (Other); University of Minnesota (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Vernon Michael Chinchilli, Distinguished Professor, Milton S. Hershey Medical Center
Other Study IDs: STUDY00015937; R01DK138060 (NIH); U01DK127384 (NIH)
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Pancreatitis
Keywords: Diabetes; Continuous Glucose Monitoring
MeSH Terms: conditions — Pancreatitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CGM: Continuous Glucose Monitoring (CGM)
  Interventions: Device: Dexcom Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Dexcom Continuous Glucose Monitor (CGM) — Dexcom Continuous Glucose Monitor which measures and records a participant's serum glucose level

SUMMARY:
The DREAM-ON study will investigate whether continuous glucose monitoring (CGM) is useful to predict risk for developing diabetes mellitus (DM) and pre-diabetes mellitus (PDM), the need for insulin therapy among those who develop DM, and to determine whether CGM can provide insight into the pathophysiology and DM subtype among participants who have experienced an episode of acute pancreatitis (AP). Thus, the results of the DREAM-ON study could inform future clinical practice guidelines for the management AP as well as potentially extending the licensing authorization for CGM to include use in patients with pancreatogenic (Type 3c) DM.

DETAILED DESCRIPTION:
The primary objective of the DREAM-ON study is to determine if continuous glucose monitoring (CGM) metrics can predict the incidence of prediabetes mellitus (PDM) and diabetes mellitus (DM) after an episode of acute pancreatitis (AP). Secondary objectives of the DREAM-ON study include determining if CGM metrics predict the need for insulin therapy in participants who develop diabetes mellitus after AP, and if CGM metrics correlate with measures of insulin secretion and insulin resistance.

The specific aims of the DREAM-ON study are as follows:

Aim 1: To test whether standard CGM metrics predict incident DM. The investigators will perform blinded CGM in DREAM-ON participants at their scheduled visits at months 3, 12, 24 and subsequent annual visits. The investigators will test whether standard CGM metrics (mean glucose, time in tight range 70-140, time in range 70-180, time above 180 mg/dL, time above 250 mg/dL and glucose CV) predict incident DM determined by fasting plasma glucose (FPG), HbA1c, oral glucose tolerance testing (OGTT) and clinical report.

Aim 2: To test whether CGM metrics predict need for insulin therapy in patients who develop DM after AP. From blinded CGM, we will test whether standard CGM metrics (mean glucose, time in tight range 70-140, time in range 70-180, time above 180 mg/dL, time above 250 mg/dL and glucose CV) as well as other indices of glucose variability, including mean amplitude of glycemic excursions (MAGE), predict need for long-term insulin therapy.

Aim 3: To determine whether CGM metrics correlate with measures of insulin secretion and insulin resistance. The investigators will test whether standard and advanced CGM metrics correlate with measures of insulin secretion and insulin resistance derived from the OGTT, the mixed meal tolerance test (MMT) and the frequently sampled intravenous glucose tolerance test (FSIGTT). The investigators also will test whether these metrics can be used as a surrogate to predict diabetes subtype (i.e., insulin deficient vs. insulin resistant).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute pancreatitis (AP) 0-90 days prior to enrollment
* Participant fully understands and is able to participate in all aspects of the study, including providing informed consent, completion of case report forms, telephone interviews, metabolic testing, and planned longitudinal follow-ups

Exclusion Criteria:

* Diagnosis of definite chronic pancreatitis (CP) at enrollment (see also study definitions) based on either of the following criteria met by computed tomography (CT) scan (including non-contrast enhanced) or Magnetic Resonance Imaging (MRI) or Magnetic Resonance Cholangiopancreatography (MRCP): (a) Parenchymal or ductal calcifications on CT scan (after excluding the possibility that calcifications are vascular); (b) Intraductal filling defects suggestive of calcifications on MRI and/or MRCP
* Potential participants with post-endoscopic retrograde cholangiopancreatography (ERCP) AP who are hospitalized for <48 hours.
* Prior (i.e., before enrollment) direct endoscopic necrosectomy of the pancreas or percutaneous necrosectomy or drainage of necrotic collection(s). Participants who require this during follow-up will remain in the study
* Pancreatic tumors, including ductal adenocarcinoma, neuroendocrine tumors, and metastasis
* Confirmed or suspected cystic tumor associated with main pancreatic duct dilation, or believed to be the cause of AP (in the site-PI's judgement).
* Prior pancreatic surgery, including, but not limited to: distal pancreatectomy, pancreaticoduodenectomy, pancreatic necrosectomy, Frey procedure.
* Use of disallowed concomitant medications within 30 days prior to enrollment. A comprehensive list of disallowed medications will be included and routinely updated in the study's Manual of Procedures
* Severe systemic illness that in the judgement of the investigative team will confound outcome assessments of diabetes mellitus and immunological outcomes or pose additional risk for harms, including: history of solid organ transplant, acquired immunodeficiency syndrome (AIDS), active treatment for cancer (except non-melanoma skin cancer) within 12 months prior to enrollment, chronic kidney disease with estimated glomerular filtration rate (eGFR) < 30 or on dialysis prior to AP, and decompensated cirrhosis (based on imaging or biopsy), or any other medical condition that in the opinion of the site-PI carries a life expectancy of <12 months
* Known pregnancy at the time of enrollment. Participants who become pregnant during follow-up will remain in the study, but may have modified study assessments for safety as detailed in the Manual of Procedures
* Incarceration
* Any other condition or factor that would compromise the participant's safety or the scientific integrity of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
pre-diabetes mellitus following an episode of acute pancreatitis | any time during the 36-month longitudinal follow-up period
  time to onset of pre-diabetes mellitus during the 36-month longitudinal follow-up period
diabetes mellitus following an episode of acute pancreatitis | any time during the 36-month longitudinal follow-up period
  time to onset of diabetes mellitus during the 36-month longitudinal follow-up period

SECONDARY OUTCOMES:
initiation of insulin therapy | any time during the 36-month longitudinal follow-up period
  time to onset of the initiation of insulin therapy of any type (basal, mixed, prandial, basal/bolus) for two or more weeks in a non-hospitalized setting after developing diabetes mellitus
insulin secretion | during the oral glucose tolerance test (OGTT) administered at 3, 12, 24, and 36 months
  insulin secretion during the oral glucose tolerance test (OGTT)
insulin sensitivity | during the oral glucose tolerance test (OGTT) administered at 3, 12, 24, and 36 months
  insulin sensitivity during the oral glucose tolerance test (OGTT)
fasting glucose | during the mixed meal tolerance test (MMTT) administered at 3, 12, 24, and 36 months
  fasting glucose during the mixed meal tolerance test (MMTT)
peak value glucose | during the mixed meal tolerance test (MMTT) administered at 3, 12, 24, and 36 months
  peak value glucose during the mixed meal tolerance test (MMTT)
meal-stimulated insulin | during the mixed meal tolerance test (MMTT) administered at 3, 12, 24, and 36 months
  meal-stimulated insulin during the mixed meal tolerance test (MMTT)
acute insulin response to glucose | during the frequently sampled intravenous glucose tolerance test (FSIGTT) administered at 3 and 12 months
  acute insulin response to glucose during the frequently samples intravenous glucose tolerance test (FSIGTT)

CONTACTS AND LOCATIONS:
Overall Officials: Vernon M Chinchilli, PhD, Principal Investigator — Penn State College of Medicine; Richard E Pratley, MD, Principal Investigator — AdventHealth
Locations (13):
- United States (13):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - AdventHealth, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data from final locked datasets will be made available to other researchers outside the DREAM-ON investigative team. The plan for data sharing incorporates a strategy that recognizes the importance of protecting participants' rights to individual privacy and is compliant with HIPAA regulations and NIH requirements (https://grants.nih.gov/grants/policy/data_sharing).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available one year after publication of the primary manuscript of the DREAM-ON manuscript. The data will be available indefinitely at the NIDDK Central Repository.
Access Criteria: Instructions for requesting data from the NIDDK Central Repository appear at the following web site: https://repository.niddk.nih.gov/pages/overall_instructions/
URL: https://repository.niddk.nih.gov/home/